CLINICAL TRIAL: NCT01428063
Title: An Open-Label Re-Treatment Study With PegInterferon Alfa-2a, Ribavirin and BMS-790052 With or Without BMS-650032 for Subjects With Chronic Hepatitis C
Brief Title: Study of pegInterferon Alfa-2a, Ribavirin, and Daclatasvir (BMS-790052) With or Without BMS-650032 for Participants in Some Hepatitis C Virus Trials
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-026; 2011-000836-27 (EudraCT Number)
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daclatasvir + Asunaprevir + PegIFNα-2a + Ribavirin (Experimental): Patients received daclatasvir, 60-mg tablet, by mouth once daily + asunaprevir, 100-mg capsule or 200-mg tablet, by mouth twice daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin
- Daclatasvir + PegIFNα-2a + Ribavirin (Experimental): Patients received daclatasvir, (two 30-mg tablets or one 60-mg tablet, by mouth once daily) + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks
  Interventions: Drug: Daclatasvir; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin
- Daclatasvir + Asunaprevir (Experimental): Patients received daclatasvir, 60-mg tablet, by mouth once daily + asunaprevir, 100-mg capsule, by mouth twice daily for 24 weeks
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Asunaprevir
  Other Names: BMS-650032
  Arms: Daclatasvir + Asunaprevir; Daclatasvir + Asunaprevir + PegIFNα-2a + Ribavirin
Drug: Pegylated interferon alfa-2a
  Other Names: pegIFNα-2a, Pegasys®
  Arms: Daclatasvir + Asunaprevir + PegIFNα-2a + Ribavirin; Daclatasvir + PegIFNα-2a + Ribavirin
Drug: Ribavirin
  Other Names: Copegus®
  Arms: Daclatasvir + Asunaprevir + PegIFNα-2a + Ribavirin; Daclatasvir + PegIFNα-2a + Ribavirin

SUMMARY:
The purpose of this study is to provide anti-hepatitis C virus drugs to patients who received placebo + peginterferon alfa-2a + ribavirin in prior Bristol-Myers Squibb (BMS) studies and determine whether addition of these drugs results in higher cure rates in patients who previously failed therapy. Approximately 100 genotype 1b patients who received placebo in BMS study NCT01428063 (AI447-028) will receive active drugs in this study.

DETAILED DESCRIPTION:
* Intervention Model:

  * Parallel: for all patients entering the trial
  * Cross-over: for genotype 1b patients rolling over from NCT01428063 (AI447-028) who require rescue therapy after initial treatment in this study
* Peginterferon alfa-2a
* Ribavirin
* Daclatasvir
* Asunaprevir

ELIGIBILITY:
Key Inclusion Criteria:

* Prior participation in any BMS-790052, BMS-650032, or BMS-791325 trial and assigned to control arm (pegIFNα-2a/ribavirin + placebo) during the trial
* Hepatitis C virus (HCV) genotype 1, 2, 3, or 4 (mixed genotypes are not permitted)
* HCV RNA viral load detectable

Key Exclusion Criteria:

* Discontinuation from a prior BMS HCV clinical trial due to a pegIFNα-2a/ribavirin-related event
* Any anti-HCV therapy following initial treatment with BMS-650032, BMS-790052, or BMS-791325
* Positive for hepatitis B infection (hepatitis B surface antigen) or HIV-1 or HIV-2 antibody at screening
* Evidence of medical condition associated with chronic liver disease other than HCV infection
* Evidence of decompensated cirrhosis based on radiologic criteria or biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (87):
- United States (20):
  - Baptist Medical Center South, Montgomery, Alabama
  - Scripps Clinic, La Jolla, California
  - Scpmg/ Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University Of Colorado Denver And Hospital, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Uf Hepatology Research At Ctrb, Gainesville, Florida
  - Schiff Center For Liver Diseases, Miami, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, P.A., Catonsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - North Shore Long Island Jewish Health System, Manhasset, New York
  - Duke University Medical Center, Durham, North Carolina
  - Options Health Research, Llc, Tulsa, Oklahoma
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Baylor College Of Medicine, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Dean Clinic, Madison, Wisconsin
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Prov. Buenos Aires, Buenos Aires
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- Australia (10):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Fremantle, Western Australia
  - Local Institution, Perth, Western Australia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Canada (6):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Vaughan, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Local Institution, Hvidovre, Denmark
- France (12):
  - Local Institution, Bondy
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution, Villejuif
- Germany (6):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
- Local Institution, Thesaloniki, Greece
- Local Institution, Dublin, Dublin, Ireland
- Italy (8):
  - Local Institution, Brescia
  - Local Institution, Cisanello (pisa)
  - Local Institution, Messina
  - Local Institution, Milan
  - Local Institution, Pavia
  - Local Institution, Roma
  - Local Institution, Torino
  - Local Institution, Viale Del Policlinico, 155
- Local Institution, Guadalajara, Jalisco, Mexico
- Local Institution, Auckland, New Zealand
- Poland (2):
  - Local Institution, Bialystok
  - Local Institution, Wroclaw
- South Korea (4):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Local Institution, Barcelona, Spain
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm
- Taiwan (2):
  - Local Institution, Taichung
  - Local Institution, Taipei
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Glasgow, Lanarkshire

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 92 centers in 20 countries.
Pre-assignment Details: A total of 276 participants were enrolled, 228 were randomized and 227 received treatment. Participants were not treated because they no longer met study criteria (n=41), withdrew their consent (n=4), showed poor/non-compliance (n=1) or were lost to follow-up (n=2). One participant was randomized by mistake but received no treatment.
Groups:
- Daclatasvir + Asunaprevir: Participants received daclatasvir, 60-mg tablet, by mouth once daily + asunaprevir, 100-mg capsule, by mouth twice daily for 24 weeks
- Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin: Participants received daclatasvir, 60-mg tablet, by mouth once daily + asunaprevir, 100-mg capsule or 200-mg tablet, by mouth twice daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks
- Daclatasvir + pegIFN-2a+ Ribavirin: Participants received daclatasvir, 60-mg tablet, by mouth once daily + pegIFNα-2a, 180-μg solution, Participants received daclatasvir, 60-mg tablet, by mouth once daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
Period: Overall Study
Arm/Group | Daclatasvir + Asunaprevir | Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin | Daclatasvir + pegIFN-2a+ Ribavirin
Started | 99 | 122 | 6
Completed | 89 | 112 | 5
Not Completed | 10 | 10 | 1
Not completed — Lack of Efficacy | 8 | 4 | 1
Not completed — Adverse Event | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — No longer meets study criteria | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Daclatasvir + pegIFN-2a+ Ribavirin: Patients received daclatasvir, 60-mg tablet, by mouth once daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Daclatasvir + Asunaprevir | Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin | Daclatasvir + pegIFN-2a+ Ribavirin | Total
Number analyzed (Participants) | 99 | 122 | 6 | 227
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 80 | 114 | 6 | 200
  65 years and older | 19 | 8 | 0 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 84 | 2 | 134
  Male | 51 | 38 | 4 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Week 12 (SVR12) for All Nonresponders With Genotype 1 Hepatitis C Virus (HCV)
Description: SVR12 defined as HCV RNA<limit of quantitation at follow-up Week 12. Nonresponder (NR)=prior NR to pegIFN-2a or ribavirin.
Time Frame: Week 12 (Follow-up period)
Population: Participants with genotype 1 HCV who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Daclatasvir + Asunaprevir + PegIFNα-2a + Ribavirin (NR): Participants received daclatasvir, 60-mg tablet by mouth once daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly for 24 weeks + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks
Arm/Group | Daclatasvir + Asunaprevir + PegIFNα-2a + Ribavirin (NR)
Number analyzed (Participants) | 37
Percentage of participants | 94.6 [81.8 to 99.3]

2. Secondary Outcome: Percentage of Participants Other Than Genotype 1 With Sustained Virologic Response at Post Treatment Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target detected or target not detected at follow-up Week 12.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in all treated participants who did not exhibit Genotype 1. One subject with indeterminate genotype in the Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin Arm/Group was excluded from the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Daclatasvir + Asunaprevir: Participants received daclatasvir (DCV), 60 mg tablet, by mouth once daily + asunaprevir (ASV), 100 mg capsule, by mouth twice daily for 24 weeks.
- DCV + ASV + pegIFN-2a+ Ribavirin (Genotype 4): Genotype 4 participants received DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegylated interferon alfa-2a(pegIFNα2a), 80 μg solution, subcutaneously weekly + ribavirin (RBV), weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures): Participants who were nor responders to earlier DCV/pegIFN/RBV therapy were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures): Participants who were nor responders to earlier ASV/pegIFN/RBV therapy were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures): Participants who were nor responders to earlier boceprevir(BOC) /pegIFN/RBV therapy were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures): Participants who were nor responders to earlier telaprevir (TVR) /pegIFN/RBV therapy were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Treatment Naive): HCV GT-1a infection treatment-naive participants were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 12 weeks.
- DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers): pegIFNα /RBV relapsers were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 12 week.
- DCV + pegIFN-2a+ RBV: Participants received daclatasvir, 60-mg tablet, by mouth once daily + pegIFNα-2a, 180-μg solution, Participants received daclatasvir, 60-mg tablet, by mouth once daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin (Genotype 4) | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 10 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Percentage of participants | 85.9 [77.4 to 92.0] | 90.0 [55.5 to 99.7] | 40.0 [12.2 to 73.8] | 100.0 [54.1 to 100.0] | 90.9 [58.7 to 99.8] | 76.9 [46.2 to 95.0] | 84.0 [63.9 to 95.5] | 88.9 [51.8 to 99.7] | 50.0 [11.8 to 88.2]

3. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) at Post Treatment Week 4
Description: RVR was defined as the percentage of participants with hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target not detected at Week 4.
Time Frame: Week 4
Population: The analysis was performed in all treated participants defined as participants who received at least 1 dose of study therapy.
Measure: Number; unit: Percentage of participants
Groups:
- DCV + ASV + pegIFN-2a+ Ribavirin: Participants received DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegylated interferon alfa-2a(pegIFNα2a), 80 μg solution, subcutaneously weekly + ribavirin (RBV), weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures): Participants who were nor responders to earlier boceprevir(BOC)/pegIFN/RBV therapy were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures): Participants who were nor responders to earlier telaprevir (TVR)/pegIFN/RBV therapy were administered with DCV, 60 mg tablet, by mouth once daily + ASV,100 mg capsule or 200 mg tablet, by mouth twice daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- DCV + pegIFN-2a+ RBV: Participants received DCV, 60 mg tablet, by mouth once daily + pegIFNα2a, 80 μg solution, subcutaneously weekly + RBV, weight based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 48 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Percentage of participants | 72.7 | 91.7 | 70.0 | 83.3 | 90.9 | 76.9 | 76.0 | 88.9 | 83.3

4. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as the percentage of participants with hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target not detected at both weeks 4 and 12.
Time Frame: Week 4 and 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 48 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Percentage of participants | 67.7 | 87.5 | 70.0 | 83.3 | 81.8 | 76.9 | 64.0 | 88.9 | 83.3

5. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as the percentage of participants with hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target not detected at week 12.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 48 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Percentage of participants | 87.9 | 95.8 | 90.0 | 100.0 | 90.9 | 92.3 | 76.0 | 88.9 | 83.3

6. Secondary Outcome: Percentage of Participants With End of the Treatment Response (EOTR)
Description: EOTR was defined as the percentage of participants with hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target not detected at end of treatment.
Time Frame: End of the study (Week 24)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 48 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Percentage of participants | 85.9 | 97.9 | 90.0 | 100.0 | 90.9 | 92.3 | 84.0 | 88.9 | 83.3

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Post Treatment Week 24 (SVR24)
Description: SVR24 was defined as the percentage of participants with hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target detected or target not detected at follow-up week 24.
Time Frame: Week 24 (Follow-up)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 48 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Percentage of participants | 84.8 | 95.8 | 40.0 | 100.0 | 90.9 | 76.9 | 84.0 | 88.9 | 50.0

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to AEs, and Who Died During the Study
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: For AEs: Day 1 until last visit. For SAEs: Day 1 until 30 days post discontinuation of dosing or participation
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Daclatasvir + Asunaprevir | DCV + ASV + pegIFN-2a+ Ribavirin | DCV + ASV + pegIFN-2a+ RBV (Prior DCV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior ASV Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior BOC Failures) | DCV + ASV + pegIFN-2a+ RBV (Prior TVR Failures) | DCV + ASV + pegIFN-2a+ RBV (Treatment Naive) | DCV + ASV + pegIFN-2a+ RBV (pegIFNα /RBV Relapsers) | DCV + pegIFN-2a+ RBV
Number analyzed (Participants) | 99 | 48 | 10 | 6 | 11 | 13 | 25 | 9 | 6
Participants
  SAEs | 4 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
  AEs leading to discontinuation of therapy | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For AEs: From Day 1, first dose until participant's last scheduled visit. For SAEs: Date of participant's written consent until 30 days post discontinuation of dosing or participation in the study if the last scheduled visit occurred later (72 weeks).
Description: On treatment period.
Groups:
- Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin: Participants received daclatasvir, 60-mg tablet by mouth once daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly for 24 weeks + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks.
- Daclatasvir + pegIFN-2a+ Ribavirin: Participants received daclatasvir, 60-mg tablet, by mouth once daily + pegIFNα-2a, 180-μg solution, subcutaneously weekly + ribavirin, weight-based dosing (<75 kg=1000 mg once daily; >=75 kg=1200 mg once daily) for 24 weeks
Arm/Group | Daclatasvir + Asunaprevir | Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin | Daclatasvir + pegIFN-2a+ Ribavirin
Serious Adverse Events (participants affected / at risk) | 4/99 | 3/122 | 0/6
Other Adverse Events (participants affected / at risk) | 58/99 | 118/122 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Asunaprevir (N=99) | Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin (N=122) | Daclatasvir + pegIFN-2a+ Ribavirin (N=6)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Asunaprevir (N=99) | Daclatasvir + Asunaprevir + pegIFN-2a+ Ribavirin (N=122) | Daclatasvir + pegIFN-2a+ Ribavirin (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 6 | 8 | 0
Asthenia (General disorders) | 2 | 15 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 1
Influenza like illness (General disorders) | 5 | 45 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 5 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 2
Nausea (Gastrointestinal disorders) | 14 | 31 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 15 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 23 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 16 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 14 | 2
Fatigue (General disorders) | 15 | 65 | 3
Depression (Psychiatric disorders) | 0 | 6 | 1
Dry eye (Eye disorders) | 0 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 22 | 2
Dysgeusia (Nervous system disorders) | 0 | 8 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 9 | 1
Transaminases increased (Investigations) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 5 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 8 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 23 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 10 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Insomnia (Psychiatric disorders) | 3 | 25 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 14 | 2
Nasopharyngitis (Infections and infestations) | 7 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 30 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 13 | 2
Amnesia (Nervous system disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 20 | 2
Headache (Nervous system disorders) | 17 | 43 | 3
Irritability (Psychiatric disorders) | 1 | 11 | 1
Pyrexia (General disorders) | 4 | 17 | 2
Weight decreased (Investigations) | 1 | 4 | 1
Chills (General disorders) | 1 | 10 | 2
Constipation (Gastrointestinal disorders) | 5 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 33 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.